CLINICAL TRIAL: NCT04562376
Title: High-intensity Resistance Training in People With Multiple Sclerosis Experiencing Fatigue - Effects on Functioning, Wellbeing and Inflammatory Biological Markers
Brief Title: High-intensity Resistance Training in People With Multiple Sclerosis Experiencing Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Neuro+ (Industry)
Responsible Party: Principal Investigator, Marie Kierkegaard, Associate Professor (Docent), Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOR 4-2358/2020
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis; Fatigue; Exercise Therapy; Resistance Training; Cytokines
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: This is a two-armed single-blinded randomized controlled trial of high-intensity resistance training in PwMS with fatigue where one group receive training twice a week (group A) and the other group once a week (group B). The randomization procedure will be performed after baseline assessments and will be concealed and based on computer-generated block randomization with block sizes of ten. No stratification will be used. Implementation of the random allocation will be done by means of sequentially numbered sealed opaque envelops.
Who Masked: Outcomes Assessor
Masking Description: A person with no further involvement in the study will manage the randomization. A research assistant will assign participants with an identification number which will be used during baseline and follow-up assessments to ensure blinding of the assessors. Thus, outcome assessors are blinded for group allocation. Data entry will be executed by a person blinded for group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The program consists of high-intensity resistance training for 60 minutes twice a week for group A during 12 weeks at the Karolinska University Hospital under the supervision of a physiotherapist. Participants in group A will have different possible training alternatives every week to ensure availability, and they will train in groups of three to five persons/session.
  Interventions: Other: High-intensity resistance training
- Group B (Active Comparator): The program consists of high-intensity resistance training for 60 minutes once a week for group B during 12 weeks at the Karolinska University Hospital under the supervision of a physiotherapist. Participants in group B will have different possible training alternatives every week to ensure availability, and they will train in groups of three to five persons/session.
  Interventions: Other: Low frequency of high-intensity resistance training

INTERVENTIONS:
Other: High-intensity resistance training — The program consists of high-intensity resistance training for 60 minutes twice a week (group A) during 12 weeks
  Arms: Group A
Other: Low frequency of high-intensity resistance training — The program consists of high-intensity resistance training for 60 minutes once a week (group B) during 12 week
  Arms: Group B

SUMMARY:
Fatigue is one of the most frequently reported and disabling impairments in multiple sclerosis (MS) and is associated with activity limitations, participation restrictions and reduced health-related quality of life (HRQL).MS fatigue is thought to be related to the disease itself, where increased levels of inflammatory biological markers (cytokines) are contributing. Resistance training may have an anti-inflammatory effect where a higher intensity is thought to have a more profound effect. Moderate-intensity resistance training is well tolerated in people with MS (PwMS) and can reduce self-reported fatigue. There is, however, a lack of high-quality studies including only fatigued PwMS when evaluating exercise regimes. Furthermore, the optimal dose (i.e. the combination of duration, frequency and intensity) is not known. Our hypothesis is that high-intensity resistance training will have positive effects in fatigued PwMS on functioning (fatigue, mood, activities and participation) and wellbeing/HRQL; and a positive immunomodulatory effect measured by inflammatory biological markers in blood. Further, that high-intensity resistance training twice a week will be superior to once a week

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is chronic inflammatory neurodegenerative disease. About two-thirds of persons with MS (PwMS) report MS-related fatigue. It is a most disabling impairment and is associated with activity limitations, participation restrictions and reduced health-related quality of life (HRQL). MS fatigue may be related directly to the disease, e.g. inflammation. Resistance training can have direct effects on the MS disease by modulating cytokine levels, where a higher intensity is thought to have a more profound effect. Thus, there are reasons to hypothesise that high-intensity resistance training might reduce fatigue in PwMS. There are, however, no randomized controlled trials (RCTs) on resistance training in PwMS with fatigue. Although the recommendation of resistance training for adults with chronic diseases is twice a week, most primary health-care providers in Sweden only offer supervised training once a week for a limited period, e.g. 8-12 weeks. Thus, our aims are to evaluate the effects of 12 weeks high-intensity resistance training on functioning (fatigue, mood, activities and participation), wellbeing/HRQL and on inflammatory biological markers (e.g. cytokines) in blood. In this two-armed single-blinded RCT, 90 PwMS with fatigue will be recruited and randomly assigned to receive high-intensity resistance training under the supervision from a physiotherapist twice a week (group A) or once a week (group B). Primary outcome is fatigue measured with a patient reported outcome, i.e. the Fatigue Scale for Motor and Cognitive Functions (FSMC), and a change-score of ten points is considered clinically meaningful. Secondary outcomes include measures of mood, participation, self-perceived impact of MS, wellbeing/HRQL and inflammatory biological markers in blood. Data will be collected at baseline and within a week after the last training session of the 12-week intervention. All participants will after the end of intervention be offered a prescription of physical activity (FaR), and have the opportunity for follow-up telephone calls at 3-, 6- and 12 months after the end of the intervention. Assessment of fatigue will also be performed at these follow-up telephone sessions. Fatigue assessments from a natural history cohort (Combat study) will be available for comparisons of natural fluctuations of fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years with the diagnosis MS according to the revised McDonald Criteria, having fatigue (i.e. ≥ 53 FSMC sum score), able to understand and communicate in Swedish, and not practicing high-intensity training within 6 months prior to the trial.

Exclusion Criteria:

* Other conditions or diagnoses judged to potentially interfere with the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Scale for Motor and Cognitive Functions | Directly after the intervention (ie change from assessments at baseline to follow-up after the 12 week intervention)
  Fatigue measured with the FSMC, minimum value 20, maximum value 100, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Fatigue Severity Scale | Directly after intervention
  Fatigue measured with the FSS, minimum value 1, maximum value 7, higher scores mean a worse outcome
Hospital Anxiety and Depression Scale | Directly after the intervention
  Mood measured with HADS, Anxiety and depression subscales, minimum value 0, maximum value 21, higher scores mean a worse outcome
Occupational Gaps Questionnaire | Directly after the intervention
  Participation in everyday occupations measured with the OGQ, minimum value 0, maximum value 30, higher scores mean a worse outcome
Multiple Sclerosis Impact Scale-29 | Directly after the intervention
  Health-related quality of life/impact of MS measured with the MS Impact Scale-29, Physical and psychological subscales, minimum value 0, maximum value 100, higher scores mean a worse outcome
Euroqool five dimension five level | Directly after the intervention
  Wellbeing/health-related quality of life measured with the EQ-5D-5L, minimum value 0, maximum value 1, higher scores mean a better outcome
Euroqool visual analogue scale | Directly after the intervention
  Wellbeing/health-related quality of life measured with the EQ VAS, minimum value 0, maximum value 100, higher scores mean a better outcome
Multiplex proteomic immunoassay and enzyme-linked immunosorbent assay | Directly after the intervention
  Analyses of inflammatory biological markers (cytokines) in blood will be analysed, a minimum and maximum value can not be specified, and higher or lower values will have different meaning depending on which biological marker (cytokine)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Kierkegaard, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Academic Specialist Center, , Stockholm Health Services, Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in a publication, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication and ending 2 years after publication
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve the aims in the approved proposal. Proposals should be directed to marie.kierkegaard@ki.se